CLINICAL TRIAL: NCT06230653
Title: A Single-centre, Randomised, Prospective Agreement Study to Determine the Clinical Performance and Safety of a Best Practice Medical Device With a Novel Sensor
Brief Title: Mechanomyography Reloaded? A Randomized Prospective Agreement Study
Acronym: MEMORY
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Ulm (Other)
Responsible Party: Principal Investigator, Manfred Blobner, Principal Investigator, University Hospital Ulm
Other Study IDs: MEMORY
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Neuromuscular Blockade
Keywords: Mechanomyography; Neuromuscular Blockade; Electromyography; Tetanic fading

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MMG on dominant arm: Mechanomyography-device will be examined on the dominant arm.
- MMG on non-dominant arm: Mechanomyography-device will be examined on the non-dominant arm.

SUMMARY:
Neuromuscular monitoring is used to evaluate neuromuscular function intraoperatively and to ensure complete neuromuscular recovery at the end of anaesthesia. Therefore, the lack of reliable neuromuscular monitoring devices that are not cumbersome to use is a major shortcoming for anaesthesia. A recently developed mechanomyography (MMG) device may meet these partially unmet needs due to its measurement of the patient's contractile force instead of its surrogates (i.e., acceleration, velocity), including the response to physiologically relevant tetanic stimulation. However, it is unclear whether the reliability of the newly developed MMG device is similar to or better than the currently available gold standard of neuromuscular monitoring based on electromyography (EMG).

DETAILED DESCRIPTION:
The MEMORY trial is a randomized clinical agreement study which will prospectively enrol thirty ASA 1 or 2 patients ≥ 18 years scheduled for non-cardiac surgery requiring general anaesthesia and neuromuscular blockade for optimisation of surgical conditions. The patient's neuromuscular function is measured on one hand with MMG and the other hand with EMG in a randomised fashion. Additionally, randomisation will be stratified the domination of one hand.

In the MEMORY trial we will test the hypothesis, that a newly developed MMG sensor provides not less reliable measurements of neuromuscular function compared to EMG in adult patients. Reliability includes agreement, precision, and the absence of staircase phenomenon and idiosyncratic responses to train-of-four (TOF) stimulation. In addition, we will explore if measurement of tetanic fade will provide more precise information about complete neuromuscular recovery than the current standard of TOF ratio >0.9.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* ASA < 3
* scheduled for non-cardiac surgery requiring general anaesthesia and neuromuscular blockade for optimisation of surgical conditions
* positioning during surgery with intraoperative access to both arms

Exclusion Criteria:

* allergy to muscle relaxants and reversal agents
* neuromuscular disease
* procedure is scheduled outside the operating room
* need of endotracheal intubation prior to surgery
* need of rapid sequence induction
* pregnancy, breastfeeding or 30 days postpartum
* surgical procedure or examination findings which are a contraindication for a supraglottic airway device
* employee of the investigator or study site directly involved in this study or other studies under the direction of the investigator or study site
* family member of the investigator
* custodial accommodation
* alcohol or drug abuse
* patients with preceding injuries impairing muscle or nerve function of the arm
* Participation in other studies with investigational drugs or devices within 4 weeks prior to screening or missing agreement not to participate in any other study at the same time or within a period of one month after the MEMORY study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The MEMORY trial is a randomized clinical agreement study which will prospectively enrol adult ASA 1 or 2 patients scheduled for non-cardiac surgery requiring general anaesthesia and neuromuscular blockade for optimisation of surgical conditions.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-22 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Precision of the Mechanomyography | intraoperative
  Measured by the repeatability coefficient at baseline and at complete neuromuscular recovery

SECONDARY OUTCOMES:
Agreement of the TOF ratio between Electromyography and Mechanomyography | intraoperative
  Agreement of the TOF ratio at 7 predefined TOF ratios: 0.3, 0.4, 0.5, 0.6, 0.7, 0.8, and 0.9
Confirmation of handling and precision of Mechanomyography sensor | intraoperative
  Investigation of baseline stability (i.e., no staircase phenomenon of the first twitch response and the TOF ratio), occurrence and magnitude of idiosyncratic TOF ratio > 1.0 during baseline measurement, repeatability of the TOF ratio during recovery from a rocuronium induced neuromuscular blockade, and sensitivity of the TOF ratio to changing the hand position during baseline measurements.

OTHER OUTCOMES:
Tetanic fade | intraoperative
  Measurement of the tetanic fading at baseline, at a TOF ratio of 0.9 measured by EMG, at a TOF ratio of 0.95 measured by EMG, and 5 min after a bolus of 2 mg/kg sugammadex

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Blobner, MD PhD, Principal Investigator — Department of Anesthesiology and Intensive Care Medicine, Technical University of Munich, Germany

REFERENCES:
- [Derived] Scholze AS, Ulm B, Kretsch N, Jungwirth B, Blobner M, Scheffenbichler FT. A single-centre, randomised comparison of the performance and safety of a novel mechanomyography sensor with electromyography. Br J Anaesth. 2026 Jan 7:S0007-0912(25)00830-X. doi: 10.1016/j.bja.2025.10.067. Online ahead of print. PMID 41506970